CLINICAL TRIAL: NCT02536820
Title: Psychoneuroimmunology Therapy in Uncontrolled Diabetic Patients: A Quasi-experimental Study
Acronym: PNIT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Salutia (Other)
Collaborators: Coomeva E.P.S (Unknown); Sinergia (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PNIT2015
Record Dates: First submitted 2015-08-28; First posted 2015-09-01 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional treatment + PNIT (Other): PNIT: Psychoneuroimmuno therapy Conventional treatment: Usual treatment that each diabetic patient recieved
  Interventions: Behavioral: psychoneuroimmune therapy
- Conventional treatment (Active Comparator): Conventional treatment: Usual treatment that each diabetic patient recieved
  Interventions: Drug: Conventional treatment

INTERVENTIONS:
Behavioral: psychoneuroimmune therapy
  Other Names: Solarte Technique
  Arms: Conventional treatment + PNIT
Drug: Conventional treatment — Actual diabetes treatment in each participant
  Arms: Conventional treatment

SUMMARY:
The Psychoneuroimmunotherapy (PNIT) is the study, modification and implementation of the interactions between the processes of adaptive behavior, neurological, endocrine and immune.

Among its premises assuming homeostasis or physiological balance as an integrated process involving the systems above mentioned.

Additionally, among the basics theme the re-mean is introduced, ie changing the direction, the function of a concept from a negative context carry a positive meaning, so that from the PNIT no disease is seen as a problem but as a situation to solve. The patient then transmits the importance of which will come.

Primary objective:

To investigate whether patients on PNIT have a higher proportion of patients achieving disease control (<7% in glycosylated hemoglobin (HBAC1) and quality of life compared with conventional treatment patients.

Methodology:

quasi-experimental, simple blind, simple blind, parallel, phase III clinical trial The investigators will follow a group of patients with type 2 diabetes mellitus durgin three months with an interim analysis a month after receiving the intervention (two visits) During each visit a trained PNIT physician assess the effectiveness, safety and quality of life of each patient.

The investigators will include male or female patients aged 18 years-old with diabetes mellitus type II in any severity, uncontrolled (> 7% Glycosilated Haemoglobin (HbAc1)) and any treatment regimen included.

The patients are not allocated by a random process and the investigators will have a convenience sample

The investigators will perform an intention to treat analysis, patients will be analyzed according to the intervention received even if this was different from the one they were assigned.

ELIGIBILITY:
Inclusion Criteria:

* Patients who wish to participate with informed consent sign.
* Diagnosed with uncontrolled diabetes mellitus type II (> 7% of HbAc1) at least six months before starting the study
* No change in medication at least three months before starting the study.
* Participants with acceptable electrocardiographic results acceptable at the study start.

Exclusion Criteria:

* Pregnant women, or planning to become pregnant during the study period.
* History of severe liver failure.
* Participants requiring elective surgeries or other procedures requiring general anesthesia for the duration of the study.
* Participants who are participating in other clinical trials involving drugs or who have participated in another clinical trial in the last three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
glycosylated hemoglobin (HbAc1 %) | 3 months

SECONDARY OUTCOMES:
Adverse events | 3 months
Fasting Plasma Glucose (mmol/L) | 3 months
Quality of life in participants in each arm | 3 months
Follow-up lost | 3 months